CLINICAL TRIAL: NCT00596128
Title: Does Implementation of a Standard Operating Procedure for Blood Sugar Control Into Daily Clinical Routine Improve Care of Patients
Brief Title: Standard Operating Procedures in Daily Clinical Routine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Jens Scholz, Department of Anaesthesiology, UK S-H Campus Kiel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UK-SH_Hanss_2008/01
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Blood Glucose
Keywords: Blood glucose; Clinical pathways
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Blood sugar monitoring and intervention as clinical routine, no SOP defined and implemented
- 2 (Experimental): Blood sugar monitoring after implementation of SOP
  Interventions: Behavioral: Implementation of SOP

INTERVENTIONS:
Behavioral: Implementation of SOP — SOP for blood sugar monitoring and intervention will be defined and ICU nurses will be educated to use this SOP in clinical routine
  Other Names: Insulin
  Arms: 2

SUMMARY:
Primary study endpoint: blood sugar values

Patients: Patients admitted to an ICU

5 steps:

1. Routine treatment,
2. Implementation of SOP for blood sugar monitoring and intervention,
3. Education of intensive care nurses,
4. 6 months free interval without further education or check-up of SOP implementation,
5. Check of SOP implementation and clinical outcome concerning range of blood sugar

DETAILED DESCRIPTION:
SOP for blood glucose monitoring and treatment was implemented on an intensive care unit. Staff was trained. After a free interval patient's outcome was monitored in terms of daily blood sugar profile prior implementation of SOP and after implementation+free interval of SOP.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an ICU

Exclusion Criteria:

* Patient's or close relative's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
blood sugar range | 4 times a day for total ICU stay

SECONDARY OUTCOMES:
ICU length of stay | After discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: jens Scholz, MD, Chair, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, UK S-H Campus Kiel, kiel, Germany
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, UK S-H Campus Kiel, Kiel, Schleswig-Holstein, Germany